CLINICAL TRIAL: NCT02095860
Title: An Open-label, Randomized, Crossover Study to Assess the Effect of Food on the Pharmacokinetics of Daclatasvir, Asunaprevir, and BMS-791325 Following Administration of a Single Fixed Dose Combination of DCV 3DAA FDC in Healthy Subjects
Brief Title: Food Effect of a Fixed Dose Combination of Daclatasvir, Asunaprevir and BMS-791325
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: AI443-111
Record Dates: First submitted 2014-03-21; First posted 2014-03-26 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A: DCV 3DAA FDC fasted state (Experimental): DCV 3 Direct Acting Antiviral (DAA) Fixed Dose Combination (FDC) tablet by mouth once on specified days in fasted state
  Interventions: Drug: DCV 3DAA FDC
- Treatment B: DCV 3DAA FDC with high-fat meal (Experimental): DCV 3DAA FDC tablet by mouth once on specified days with high-fat meal
  Interventions: Drug: DCV 3DAA FDC
- Treatment C: DCV 3DAA FDC with light meal (Experimental): DCV 3DAA FDC tablet by mouth once on specified days with light meal
  Interventions: Drug: DCV 3DAA FDC

INTERVENTIONS:
Drug: DCV 3DAA FDC — Fixed Dose Combination of Daclatasvir (DCV), Asunaprevir (ASV) and BMS-791325

SUMMARY:
The purpose of this study is to assess the effect of a high fat meal and light meal on the blood levels of Daclatasvir, Asunaprevir and BMS-791325 after administration of the 3 drugs as a fixed-dose combination in healthy subjects.

DETAILED DESCRIPTION:
IND Number: 100,932/79,599/101,943

Primary Purpose:

Other: Phase 1 clinical pharmacology bioavailability study to assess food effect

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Healthy male and female subjects ages 18 to 49 years, inclusive.
* Women of childbearing potential must be using an acceptable method of contraception for at least 4 weeks prior to study drug administration.

Exclusion Criteria:

* Any significant acute or chronic medical illness
* Current or recent (within 3 months of study drug administration) gastrointestinal disease
* Any gastrointestinal surgery that could impact upon the absorption of study drug, including cholecystectomy
* History of biliary disorders, including Gilbert's syndrome or Dubin-Johnson disease
* Use of tobacco-containing or nicotine-containing products
* Any of the following on 12-lead electrocardiogram (ECG) prior to study drug administration, confirmed by repeat:

  * PR ≥210 msec
  * QRS ≥120 msec
  * QT ≥500 msec
  * QTcF ≥450 msec
* Any of the following laboratory results outside of the ranges specified below prior to study drug administration, confirmed by repeat:

  * Alanine aminotransferase (ALT) >Upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) >ULN
  * Total bilirubin (TBILI) >ULN
  * Creatinine >ULN

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of DCV, ASV and BMS-791325 | Day 1 to Day 13
Area under the plasma concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] of DCV, ASV and BMS-791325 | Day 1 to Day 13

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration [AUC(0-T)] for DCV, ASV and BMS-791325 | Day 1 to Day 13
Time of maximum observed plasma concentration (Tmax) for DCV, ASV and BMS-791325 | Day 1 to Day 13
Terminal plasma half life (T-HALF) for DCV, ASV and BMS-791325 | Day 1 to Day 13
AUC(0-T) for BMS-794712 | Day 1 to Day 13
AUC(INF) for BMS-794712 | Day 1 to Day 13
Cmax for BMS-794712 | Day 1 to Day 13
Tmax for BMS-794712 | Day 1 to Day 13
T-HALF for BMS-794712 | Day 1 to Day 13
Safety measured by incidence of adverse event (AEs), serious AEs (SAEs) and AEs leading to discontinuation | Day 1 to Day 13
Safety measured by abnormalities in vital sign measurements | Day 1 to Day 13
Safety measured by findings on electrocardiograms (ECG) measurements and physical examinations | Day 1 to Day 13
Safety measured by marked abnormalities in clinical laboratory test results | Day 1 to Day 13

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Healthcare Discoveries, Llc D/B/A Icon Development Solutions, San Antonio, Texas, United States

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx